CLINICAL TRIAL: NCT02886455
Title: Evaluation of the Influence of Output on Skin Covered by Newly Developed Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_04
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 4 (Experimental): This is a sub-study testing the effect of real output applied under two adhesive strips on the skin at two different time points (4 and 24 hours).
  There are two visits:
  Visit 1:
  Two adhesive strips (standard adhesive strip and new adhesive strip)contaminated with the subjects own output are applied on the peristomal skin and allowed to sit for 4 hours before being removed
  Visit 2: Two adhesive strips (standard adhesive strip and new adhesive strip)contaminated with the subjects own output are applied on the peristomal skin and allowed to sit for 24 hours before being removed
  Interventions: Other: Standard adhesive strip; Other: New adhesive strip

INTERVENTIONS:
Other: Standard adhesive strip — This is a standard adhesive strip (hydrocolloid)
Other: New adhesive strip — This a newly developed adhesive strip.

SUMMARY:
The study investigates the impact real output has on peristomal skin covered by a newly developed adhesive and a standard adhesive.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 4-24 hours
  The condition of the skin (transepidermal water loss) is measured after removing the adhesive by TE

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, Msc, Principal Investigator — R&D scientist
Locations (1):
- Coloplast A/S, Humlebæk, Denmark